CLINICAL TRIAL: NCT03549013
Title: The Long-Term Outcome of 3D-CT-guided Percutaneous Radiofrequency Thermocoagulation for Tumor-related Trigeminal Neuralgia: A Retrospective Study.
Brief Title: 3D-CT-guided Percutaneous Radiofrequency Thermocoagulation for Tumor-related Trigeminal Neuralgia
Status: Completed | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Fang Luo, vice director of Department of Anesthesiology and Pain Management, Beijing Tiantan Hospital
Other Study IDs: KY 2018-024-02
Record Dates: First submitted 2018-05-21; First posted 2018-06-07 (Actual); Last update posted 2018-06-07 (Actual); Status verified 2018-06

CONDITIONS: Trigeminal Neuralgia, Secondary
Keywords: Tumor-related Trigeminal Neuralgia; Percutaneous Radiofrequency Thermocoagulation; Three-dimensional Computed Tomography
MeSH Terms: conditions — Trigeminal Neuralgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is designed to investigate the effectiveness and safety of 3D-CT-guided percutaneous radiofrequency thermocoagulation for the treatment of tumor-related trigeminal neuralgia.

DETAILED DESCRIPTION:
Approximately 1-13% of trigeminal neuralgia cases are secondary to intracranial tumors, and this condition is referred to as tumor-related trigeminal neuralgia (TRTN). TRTN can result from a lesion affecting any location along the pathway of the trigeminal nerve, such as Meckel's Cave, the posterior fossa, and the cerebellopontine angle. The posterior fossa is the most common location of TRTN, whereas meningioma and epidermoid cysts are the most common pathologies. The goals of TRTN treatment include controlling tumors and relieving pain. Tumor resection is regarded as the most effective treatment, and complete tumor removal is often followed by complete pain remission. However, for patients who cannot undergo the risk of a craniotomy and those with end-stage of malignant tumors or slow-growing benign tumors, surgery may not be the best choice. Conservatively, medication is considered the first-line therapy for relieving pain. However, pharmacology cannot provide satisfactory relief for all patients, and some patients may experience intolerable side effects. For these patients, minimally invasive interventional techniques are preferred. Radiosurgery has been commonly performed for the treatment of TRTN with promising efficacy. However, this intervention is associated with delayed latency of response. Percutaneous radiofrequency thermocoagulation (PRFT) is a low-risk, minimally invasive technique with an acute success rate of 97.6-99%. PRFT remains the most common percutaneous treatment for TN. In addition, this popular procedure may also safely and effectively be repeated if pain recurs. The PRFT procedure involves positioning the radiofrequency (RF) needle at the Gasserian ganglion via the foremen ovale. Suboptimal piercing may lead to unpleasant complications, including cerebrospinal fluid leakage, cranial nerve (VI) palsy and intracranial hemorrhage. Recently, computed tomography (CT) has been demonstrated to be a useful method to identify the optimal position and predict the intraoperative difficulties of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* age>18 years,
* typical TN symptoms in the same lateral as intracranial tumors,
* uncontrolled symptoms or intolerable side effects of medication,
* pain duration longer than 90 days
* brain magnetic resonance imaging (MRI)confirmed that the trigeminal pain was secondary to intracranial tumors.

Exclusion Criteria:

* patients with infection at the puncture site,
* coagulopathy,
* epilepsy,
* other causes of TN,
* a history of mental disorders or anesthetic drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This retrospective study was conducted in Beijing Tiantan Hospital between March 2007 and February 2018. The local ethics committee approved this study and exempted the informed consent before the collection of patient data. We enrolled a total of 38 patients who fulfilled all following criteria: age>18 years; typical TN symptoms in the same lateral as intracranial tumors; uncontrolled symptoms or intolerable side effects of medication; and pain duration longer than 90 days. To confirm that the trigeminal pain was secondary to tumors, brain magnetic resonance imaging (MRI) was performed in advance. Patients with infection at the puncture site, coagulopathy, epilepsy, other causes of TN, a history of mental disorders or anesthetic drug abuse were excluded from this study.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2018-04-29 (Actual); Primary Completion 2018-05-05 (Actual); Study Completion 2018-05-05 (Actual)

PRIMARY OUTCOMES:
Cumulative recurrence-free rate | The enrollment of our study began on March 1st 2007 and ended on 31st October 2017. All following-up has been finished before February 28th 2018.
  The modified Barrow Neurological Institute (BNI) pain intensity score will be used to assess pain degree. Pain relief degree will be evaluated as BNI I= no pain without medication, BNI II= occasional pain, not require medication, BNI IIIa= no pain with medication, BNI IIIb= Controlled pain with medication, BNI IV= improved pain that inadequately controlled by medication, BNI IV= persistent pain that inadequately controlled by medication. A BNI grade that increased to IV-V from I-IIIb after operation was defined as recurrence.

SECONDARY OUTCOMES:
Patient satisfaction | From pre-operation to 1 week after operation
  Patient satisfaction is evaluated by a 5-point Likert scale, while 1 point represents very unsatisfactory and 5 points indicates very satisfactory
Adverse events | The enrollment of our study began on March 1st 2007 and ended on 31st October 2017. All following-up has been finished before February 28th 2018.
  Data regarding intra-and post=operative adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Fang Luo, M.D., Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kim SK, Kim DG, Se YB, Kim JW, Kim YH, Chung HT, Paek SH. Gamma Knife surgery for tumor-related trigeminal neuralgia: targeting both the tumor and the trigeminal root exit zone in a single session. J Neurosurg. 2016 Oct;125(4):838-844. doi: 10.3171/2015.7.JNS15451. Epub 2016 Jan 22. PMID 26799302
- [Background] Cho KR, Lee MH, Im YS, Kong DS, Seol HJ, Nam DH, Lee JI. Gamma knife radiosurgery for trigeminal neuralgia secondary to benign lesions. Headache. 2016 May;56(5):883-889. doi: 10.1111/head.12801. Epub 2016 Apr 4. PMID 27041354
- [Background] Furtado SV, Hegde AS. Trigeminal Neuralgia Due to a Small Meckel's Cave Epidermoid Tumor: Surgery Using an Extradural Corridor. Skull Base. 2009 Sep;19(5):353-7. doi: 10.1055/s-0029-1220201. PMID 20190946
- [Background] Cheng TM, Cascino TL, Onofrio BM. Comprehensive study of diagnosis and treatment of trigeminal neuralgia secondary to tumors. Neurology. 1993 Nov;43(11):2298-302. doi: 10.1212/wnl.43.11.2298. PMID 8232946
- [Background] Khan N, Michael A, Choucair A, Bit-Ivan E. Trigeminal Ganglioneuroma: A Rare Case of Trigeminal Neuralgia Caused by Cerebellopontine Angle Tumor. World Neurosurg. 2017 Mar;99:811.e7-811.e10. doi: 10.1016/j.wneu.2016.12.085. Epub 2016 Dec 30. PMID 28043883
- [Background] Kobata H, Kondo A, Iwasaki K. Cerebellopontine angle epidermoids presenting with cranial nerve hyperactive dysfunction: pathogenesis and long-term surgical results in 30 patients. Neurosurgery. 2002 Feb;50(2):276-85; discussion 285-6. doi: 10.1097/00006123-200202000-00008. PMID 11844262
- [Background] Kanpolat Y, Savas A, Bekar A, Berk C. Percutaneous controlled radiofrequency trigeminal rhizotomy for the treatment of idiopathic trigeminal neuralgia: 25-year experience with 1,600 patients. Neurosurgery. 2001 Mar;48(3):524-32; discussion 532-4. doi: 10.1097/00006123-200103000-00013. PMID 11270542
- [Background] Fraioli B, Esposito V, Guidetti B, Cruccu G, Manfredi M. Treatment of trigeminal neuralgia by thermocoagulation, glycerolization, and percutaneous compression of the gasserian ganglion and/or retrogasserian rootlets: long-term results and therapeutic protocol. Neurosurgery. 1989 Feb;24(2):239-45. doi: 10.1227/00006123-198902000-00014. PMID 2783993
- [Background] Emril DR, Ho KY. Treatment of trigeminal neuralgia: role of radiofrequency ablation. J Pain Res. 2010 Dec 12;3:249-54. doi: 10.2147/JPR.S14455. PMID 21311718